CLINICAL TRIAL: NCT02154477
Title: Effect of Intranasal Insulin on LH Concentrations in Man
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: L14-075
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: hypogonadotropic hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diabetes (Active Comparator): All patient will receive insulin at one visit and saline at another visit
  Interventions: Drug: intranasal insulin; Drug: placebo (intranasal saline)
- control (Active Comparator): All patient will receive insulin at one visit and saline at another visit
  Interventions: Drug: intranasal insulin; Drug: placebo (intranasal saline)

INTERVENTIONS:
Drug: intranasal insulin — insulin
Drug: placebo (intranasal saline) — saline

SUMMARY:
Over the last few years, studies have shown that men with type 2 diabetes sometimes develop a condition called hypogonadotrophic hypogonadism (HH). People with this condition produce little or no sex hormones. Obesity and metabolic syndrome are also associated with HH. Research suggests that insulin in the brain may benefit the glands that release these hormones. During this study, subjects will spray a small amount of insulin into their nose.This will increase insulin concentrations in the brain. The purpose of this study is to find out the effect of one dose of intranasal insulin on release of LH (a sex hormone) in obese diabetic men with HH.

DETAILED DESCRIPTION:
Studies over the last few years have clearly established that at least 25% of men with type 2 diabetes have subnormal free testosterone (T) concentrations in association with inappropriately low leutinizing hormone (LH) and FSH (follicle stimulating hormone) concentrations. These patients thus suffer from hypogonadotrophic hypogonadism (HH). Obesity and metabolic syndrome are also associated with HH. Animal studies and in vitro data have shown that insulin action and insulin responsiveness in the brain are necessary for the maintenance of the functional integrity of the hypothalamo-hypophyseal-gonadal axis. Insulin concentrations can be increased in the brain by delivering insulin intranasally with vianase device. The aim of this project is to study the effect of one dose of intranasal insulin on release of LH in obese diabetic men with HH. 15 obese men with type 2 diabetes and low free T along with normal LH concentrations will be recruited for the study. The study will be carried out at the clinical center of Texas Tech (Odessa campus). There will be two study visits, each comprising of blood tests every 15 minutes over 6 hours. 40 IU of intranasal insulin or saline will be given after a baseline period of blood sampling of 2 hours. Student's t-test will be used to compare the change in LH concentrations after intranasal saline or insulin.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18 to 75 years
* Obesity (BMI ≥30 kg/m2)
* Type 2 diabetes
* Hypogonadotropic hypogonadism defined as calculated free testosterone concentrations below 7 ng/dl along with normal or low LH concentrations

Exclusion Criteria:

* HbA1c>8.5%
* Use of preprandial insulin therapy
* Use of testosterone currently or in the past 4 months
* Use of over the counter health supplements which contain androgens
* Use of corticosteroids or narcotics in the past 3 months
* Coronary event or procedure(myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous twelve weeks
* Type I Diabetes
* Currently suffering from foot ulcer, significant periodontal disease or any other chronic infectious or inflammatory condition
* Hepatic disease (transaminase > 3 times normal) or cirrhosis
* Renal impairment (defined as glomerular filtration rate<30)
* HIV or Hepatitis C positive status
* Any other life-threatening, non-cardiac disease
* History of untreated severe obstructive sleep apnea(defined as apnea-hypopnea index ≥30)
* currently suffering from symptomatic depression, with or without treatment
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Participation in any other concurrent clinical trial
* Pituitary tumor/damage/ other trophic hormone deficiency

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MD, Principal Investigator — TTUHSC
Locations (1):
- TTTUHSC-Permian Basin, Odessa, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dhindsa S, Chemitiganti R, Ghanim H, Santiago E, Haider A, Chaar N, Mok M, McKee A, Dandona P. Intranasal Insulin Administration Does Not Affect LH Concentrations in Men with Diabetes. Int J Endocrinol. 2018 Oct 31;2018:6170154. doi: 10.1155/2018/6170154. eCollection 2018. PMID 30515210

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: lean healthy men, randomized to receive saline or insulin at first visit and the alternate treatment at second visit
- Diabetes: men with diabetes, randomized to receive saline or insulin at first visit and the alternate treatment at second visit
Period: Overall Study
Arm/Group | Control | Diabetes
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diabetes: All patients will be randomized to receive either insulin or saline at first visit and alternate treatment at the second visit
  intranasal insulin
  placebo (intranasal saline)
- Control: All control subjects will be randomized to receive either insulin or saline at first visit and alternate treatment at the second visit
  intranasal insulin
  placebo (intranasal saline)
- Total: Total of all reporting groups
Arm/Group | Diabetes | Control | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7) | 30 (9) | 48 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: LH
Description: Luteinizing hormone (LH) concentrations after intranasal insulin as compared to placebo (intranasal saline). This endpoint was measured in both arms
Time Frame: 4 hours
Population: diabetes
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Diabetes: All patient will receive insulin at one visit and saline at another visit
  intranasal insulin
  placebo (intranasal saline)
- Control: lean healthy men. All men will receive insulin at one visit and saline at the other.
Arm/Group | Diabetes | Control
Number analyzed (Participants) | 8 | 6
IU/L
  baseline | 7.7 (3) | 3.3 (1.4)
  post-intervention saline | 7.9 (4.3) | 3.8 (1.4)
  post-intervention insulin | 8 (3.4) | 3.4 (1.2)

ADVERSE EVENTS:
Time Frame: 4 hours
Description: hypoglycemia
Groups:
- Diabetes: All diabetes patients were randomized to receive either insulin or saline at one visit and the alternate treatment at the second visit.
  intranasal insulin
  placebo (intranasal saline)
- Control: All control subjects were randomized to receive either insulin or saline at one visit and the alternate treatment at the second visit.
  intranasal insulin
  placebo (intranasal saline)
Arm/Group | Diabetes | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT02154477/Prot_SAP_000.pdf